CLINICAL TRIAL: NCT06776458
Title: Beyond Cardiotoxicity: Characterizing the Long-term Cardiovascular Side Effects of Breast Cancer Endocrine Treatment
Brief Title: Chronic Impacts of Endocrine Therapy on Cardiovascular and Brain Health Outcomes in Breast Cancer
Acronym: STRIVE-Chronic
Status: Recruiting | Type: Observational
Sponsor: University of Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Cancer Research Society (Other)
Responsible Party: Principal Investigator, Amy Kirkham, Assistant Professor, University of Toronto
Other Study IDs: REB #46819
Record Dates: First submitted 2024-12-30; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer Females
Keywords: Aromatase Inhibitors; Breast Cancer Females; Heart Disease Risk Factors

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Participant blood samples will be collected, analyzed, and stored according to study protocol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (6):
- Aromatase Inhibitors (1 year): Breast cancer patients at 1-year post-diagnosis, who were treated with aromatase inhibitors
  Interventions: Other: N/A - Usual Care
- Aromatase Inhibitors (5 year): Breast cancer patients at 5-year post-diagnosis, who were treated with aromatase inhibitors
  Interventions: Other: N/A - Usual Care
- Aromatase Inhibitors (10 years): Breast cancer patients at 10-years post-diagnosis, who were treated with aromatase inhibitors
  Interventions: Other: N/A - Usual Care
- Matched Controls (1 year): A woman without a history of cancer will be recruited to match each breast cancer patient will be matched on age and BMI (within 3 years and 3 kg/m2, whenever possible)
- Matched Controls (5 years): A woman without a history of cancer will be recruited to match each breast cancer patient will be matched on age and BMI (within 3 years and 3 kg/m2, whenever possible)
- Matched Controls (10 years): A woman without a history of cancer will be recruited to match each breast cancer patient will be matched on age and BMI (within 3 years and 3 kg/m2, whenever possible)

INTERVENTIONS:
Other: N/A - Usual Care — Breast cancer survivors will have received usual care aromatase inhibitors for up to 10 years post-diagnosis.
  Groups: Aromatase Inhibitors (1 year); Aromatase Inhibitors (10 years); Aromatase Inhibitors (5 year)

SUMMARY:
Aromatase inhibitors are the most used endocrine therapy for hormone-positive breast cancer. Despite the evidence that aromatase inhibitor therapy is associated with increased risk of cardiovascular events, potentially related to the duration of use, no studies have been conducted to characterize the long-term effects of aromatase inhibitor therapy on the heart or vessel structure and function as underlying determinants of cardiovascular mortality. This study will characterize the long-term effects of aromatase inhibitor therapy on established and novel health indices for CVD in breast cancer patients, by examining cross-sectionally compare health indices 1-, 5- and 10-years post-diagnosis in breast cancer survivors to controls. Specifically, our objectives are as follows:

1. To examine the effects of aromatase inhibitor therapy on early risk indicators for cardiovascular disease in the peripheral vasculature and heart, including aortic stiffness (primary outcome) and secondary outcomes of peripheral and carotid artery stiffness, blood biomarkers (lipids), blood pressure, carotid intima media thickness, endothelial function, and left ventricular ejection fraction, global longitudinal strain, and left ventricular diastolic function, in breast cancer survivors compared to controls.
2. To examine the effects of aromatase inhibitor therapy on factors related to cerebrovascular health, autonomic regulation, and cognitive function, including BDNF, heart rate variability, cerebrovascular function in response to a supine-sit-stand maneuver and squatting challenge, and a core battery of cognitive function tests, in breast cancer survivors compared to controls.
3. To examine the effects of aromatase inhibitor therapy on body composition, bone mineral density, and protein metabolism, in breast cancer survivors compared to controls.
4. To examine the effects of aromatase inhibitor therapy on lifestyle factors (behavioural), including diet, physical activity (including cardiorespiratory fitness), sleep, stress, and quality of life, in breast cancer survivors compared to controls.

The investigators hypothesize that biologic and behavioural cardiovascular health indices will be deteriorated relative to controls as early as 1 year post-diagnosis and that prolonged use will further accelerate aging-related impairments.

ELIGIBILITY:
Inclusion Criteria:

Case group:

* Biologically female
* Post-menopausal with natural (no bilateral oophorectomy) amenorrhea for at least 1 year
* If using hormone replacement therapy, limit of a maximum of 3 years of treatment but not within the last 6 months.
* Diagnosis of stage I, II, or III breast cancer
* Hormone receptor positive breast cancer
* HER negative (ER+/PR+/HER-) breast cancer
* Breast cancer patients ~1 post-diagnosis who have received aromatase inhibitor therapy
* Breast cancer patients ~5 and ~10 years post-diagnosis who have received aromatase inhibitor therapy for at least 2 years
* Received surgery/radiation therapies

Control group:

* Biologically female
* Post-menopausal with natural (no bilateral oophorectomy) amenorrhea for at least 1 year
* If using hormone replacement therapy, limit of a maximum of 3 years of treatment but not within the last 6 months.

Exclusion Criteria:

* Previous treatment using tamoxifen endocrine therapy in a pre-or peri-menopausal setting
* Major signs or symptoms of cardiovascular diseases, diabetes, or renal disease (taken from the American College of Sports Medicine's Guidelines for Exercise Testing and Prescription 11th edition Table 2.1: pain or discomfort in the chest, neck, jaw, arms with rest or exercise, shortness of breath at rest or with mild exertion, dizziness or syncope, loss of balance or passing out, ankle edema, palpitations or tachycardia, intermittent claudication, known heart murmur, unusual fatigue with usual activities.)
* American Heart Association's absolute or relative contraindications for symptom-limited maximal exercise testing (myocardial infarction, aortic or coronary artery stenosis, heart failure, pulmonary embolism or deep vein thrombosis, inflammation of the heart (myocarditis, pericarditis, and/or endocarditis), uncontrolled cardiac arrythmia, advanced or complete electrical heart block, stroke or transient ischemia attack, blood pressure >200mmHg/100mmHg, a cancer diagnosis other than skin cancer)
* Unable to provide informed consent or communicate in English
* Mobility limitations to exercise testing (i.e., wheelchair, walker use, limp impeding walking)
* Extreme claustrophobia

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be recruited from the community in the Greater Toronto Area via posters, newsletters, social media advertisements, and word of mouth.
Sampling Method: Non-Probability Sample
Enrollment: 112 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Aortic Stiffness | Day 2 (In-Person Session)
  Aortic stiffness, measured non-invasively by pulse wave velocity, will be assessed using applanation tonometry.

SECONDARY OUTCOMES:
Brachial Artery Endothelial Function | Day 2 (In-Person Session)
  Endothelial function will be assessed using the gold standard method of flow mediated dilation (FMD) using non-invasive duplex ultrasound (GE Vivid IQ) and edge-tracking software.
Carotid Artery Stiffness | Day 2 (In-Person Session)
  Functional assessment of the carotid artery stiffness will be assessed using B-mode ultrasound and artery edge-tracking software
Carotid Intima Media Thickness | Day 2 (In-Person Session)
  Structural assessment of the carotid artery thickness will be assessed using B-mode ultrasound and artery edge-tracking software
Arterial Stiffness | Day 2 (In-Person Session)
  Measured by Pulse Wave Velocity (PWV) of the arm and leg
Left Ventricular Ejection Fraction (LVEF) | Day 2 (In-Person Session)
  Cardiac outcomes will be assessed via echocardiography (GE Vivid IQ) and analyzed using Echopac software, represented as a % using the following formula: stroke volume/end diastolic volume x 100%.
Global Longitudinal Strain | Day 2 (In-Person Session)
  Cardiac outcomes will be assessed via echocardiography (GE Vivid IQ) and analyzed using Echopac software, expressed as a percentage of the relative change in length of the left ventricle through a cardiac cycle.
Left Ventricular Diastolic Function | Day 2 (In-Person Session)
  Cardiac outcomes will be assessed via echocardiography (GE Vivid IQ) and analyzed using Echopac software, assessed by the ratio of peak early diastolic velocity to peak mitral valve velocity (E/A ratio).
Cerebrovascular Response | Day 2 (In-Person Session)
  Cerebral blood flow velocity response (delta change compared to rest) of the middle cerebral artery will be assessed using transcranial Doppler ultrasound (Neurovision Transcranial Doppler System Model 500M) in accordance with recent guidelines, in response to postural changes (sit-to-stand) and exercise (squatting).
Brain derived neurotrophic factor | Day 2 (In-Person Session)
  Brain derived neurotrophic factor will be assessed via fasted venipuncture using in-house assays.
Lipid profile | Day 2 (In-Person Session)
  HDL, LDL, total Cholesterol, Triglycerides analyzed from blood serum using a clinical assay at a core lab.
Hemoglobin A1c | Day 2 (In-Person Session)
  Analyzed from blood plasma using a clinical assay at a core lab.
Insulin resistance | Day 2 (In-Person Session)
  Calculated as Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) from fasting blood measures of glucose and insulin, analyzed using a clinical assay at a core lab.
Protein metabolism | Day 1 (At-Home Session)
  Analyzed from breathing test and urine sample before and after the participant consume a test protein drink.

OTHER OUTCOMES:
Cardiorespiratory fitness | Day 2 (In-Person Session)
  Measured as peak volume of oxygen consumption via indirect calorimetry during a cardiopulmonary exercise test on a cycle ergometer.
Framingham 10-year risk (%) | Day 2 (In-Person Session)
  Calculated using the standardized scoring system where sex-specific points are assigned to age, systolic blood pressure (dependent on treatment status), HDL, total cholesterol, smoking and diabetes status. The range for females is 0-30% where a higher score indicates a greater risk of cardiovascular disease in the next 10 years.
Heart Rate Recovery | Day 2 (In-Person Session)
  Measured as the difference between peak heart rate during the cardiorespiratory fitness test and heart rate 2-minutes into active recovery after stopping the exercise test.
Heart Rate Variability | Day 2 (In-Person Session)
  Measured as the variability in beat-to-beat heart rate during supine rest.
avO2 difference | Day 2 (In-Person Session)
  Measured by a non-invasive optical technique used to assess tissue oxygenation and hemodynamics (Near-Infrared Spectroscopy - NIRS) at rest, and during cycling exercise at ventilatory threshold, respiratory compensation point, and peak oxygen uptake.
Cardiac Output | Day 2 (In-Person Session)
  Measured continuously by a finger cuff (Finger Arterial Pressure - Finapres) at rest, and during cycling exercise at ventilatory threshold, respiratory compensation point, and peak oxygen uptake.
Stroke Volume | Day 2 (In-Person Session)
  Measured continuously by a finger cuff (Finger Arterial Pressure - Finapres) at rest, and during cycling exercise at ventilatory threshold, respiratory compensation point, and peak oxygen uptake.
Resting Blood Pressure | Day 2 (In-Person Session)
  Measured as the average of the last 5 of 6 blood pressure measurements taken 60 seconds apart using an automatic blood pressure device.
Beat-by-beat Blood Pressure | Day 2 (In-Person Session)
  Measured continuously by a finger cuff (Finger Arterial Pressure - Finapres) at rest, and during cycling exercise at ventilatory threshold, respiratory compensation point, and peak oxygen uptake.
Hemoglobin | Day 2 (In-Person Session)
  Analyzed from blood plasma using a clinical assay at a core lab.
Whole-body fat and fat-free mass | Day 2 (In-Person Session)
  Measured using a body composition device (BodPod) to estimate whole body fat (in kg and %) and fat free mass (in kg and %).
Body circumferences | Day 2 (In-Person Session)
  Circumferences of the waist, hip and neck, measured using an inelastic tape
Bone Mineral Density | Day 2 (In-Person Session)
  Assessed using a dual x-ray absorptiometry scan.
Body weight | Day 2 (In-Person Session)
  Assessed fasted in lab using a calibrated scale
Body mass index (BMI) | Day 2 (In-Person Session)
  Calculated from a measurement of height using a stadiometer and body weight (detailed above).
Dietary intake | Day 1 (At-Home Session)
  Various components of dietary intake including macronutrients and micronutrients will be assessed through 3-day food records over 2 weekdays and 1 weekend collected using ASA-24 online system.
Diet quality | Day 1 (At-Home Session)
  An overall measure of alignment with Canada's dietary guidelines measured via the Healthy Eating Food Index-2019 calculated from 3-day diet records
Depression & Anxiety | Day 1 (At-Home Session)
  Measured by the Hospital Anxiety and Depression Scale (HADS); score ranges from 0-21 for each of depression and anxiety with a higher score indicating more severe depression or anxiety
Autonomic symptoms | Day 1 (At-Home Session)
  Assessed by the COMPASS 31 (Composite Autonomic Symptom Score) questionnaire. This questionnaire provides clinically relevant scores of autonomic symptom severity. Scores range from 0 to 31 with questions in six domains: orthostatic intolerance, vasomotor, secretomotor, gastrointestinal, bladder, and pupillomotor, with a higher scoring indicating worse autonomic dysfunction.
Cognitive Function: Verbal Fluency | Day 2 (In-Person Session)
  Assessed using the Controlled Oral Word Association of the Multilingual Aphasia Exam (verbal fluency), with higher number of words produced indicative of better cognitive health.
Cognitive Function: Verbal Learning & Memory | Day 2 (In-Person Session)
  Assessed the Hopkins Verbal Learning Test (learning, memory) with an immediate recall, delayed recall, and recognition accuracy from a list of 12 words. Higher number of words are indicative of better cognitive health.
Cognitive Function: Processing Speed | Day 2 (In-Person Session)
  Assessed by the Trail Making Test (attention, speed, executive function). Shorter test time on 2 forms of the test is indicative of better cognitive health.
Cognitive Impairment | Day 2 (In-Person Session)
  Assessed by Global Deficit Score (GDS). GDS is calculated as an average score from 3 tests: 1) Hopkins Verbal Learning Test (learning, memory), 2) Trail Making Test (attention, speed, executive function), 3) Controlled Oral Word Association of the Multilingual Aphasia Exam (verbal fluency). Each subtest of the GDS has a complex scoring system, detailed above, with higher values indicating greater cognitive deficits.
Cancer-specific Quality of life (only measured in cancer group) | Day 1 (At-Home Session)
  Assessed using the Functional Assessment of Cancer Therapy - General (FACT-G), - Endocrine (FACT-ES), Cognitive (FACT-Cog) and - Fatigue (FACT-F). These are patient-reported outcome measurements used to assess health-related quality of life in patients with a history of cancer. The FACT-G is calculated from the sum of four subscales on general health related quality of life with a range of 0-108 points. The FACT-ES is a score of 19 questions with scores ranging from 0-76. The FACT-Cog contains 37 questions with a score of 0 to 132. FACT-F is calculated from the sum of 13 questions. Higher scores on each scale is indicative of better quality of life.
Musculoskeletal health | Day 1 (At-Home Session)
  Assessed using the Musculoskeletal Health Questionnaire (MSK-HQ). The MSK-HQ is a series of 15 questions with a range from 0-56 with higher scores being indicative of poorer MSK health.
Musculoskeletal pain | Day 1 (At-Home Session)
  Assessed using the Brief Pain Inventory (BPI). The BPI is scored as the average of seven pain-related questions with a range of 0-10 with higher scores representing greater pain.
Musculoskeletal osteoarthritis risk | Day 1 (At-Home Session)
  Assessed using the Western Ontario and McMaster Universities Osteoarthritis (WOMAC) Index. The WOMAC is a series of 17 questions resulting in a % (0-100) with higher scores indicative of greater osteoarthritis index.
Musculoskeletal disability | Day 1 (At-Home Session)
  Assessed using the Disabilities of the Arm, Shoulder, and Hand (DASH) Questionnaire. The DASH contains 30 questions with scores of 0 to 100 with higher scores representing higher severity in disability.
Cardiovascular risk | Day 1 (At-Home Session)
  Assessed using the INTERHEART Risk Score, a validated score for quantifying risk-factor burden without the use of laboratory testing (with higher scores indicating greater risk-factor burden).
Gender Factors | Day 1 (At-Home Session)
  Assessed by the Stanford Gender-related Variables for Health Research (GVHR) which includes questions related to seven gender-related variables: caregiver strain, work strain, independence, risk-taking, emotional intelligence, social support, and discrimination.
Health-related quality of life | Day 1 (At-Home Session)
  Assessed by RAND-36, where an independent score is provided for 8 scales ranging from 0 to 100 and 2 component summary scales ranging from 0-50 with a higher score indicating better quality of life.
Psychosocial stress | Day 1 (At-Home Session)
  Assessed by the perceived stress scale (PSS-14) where individual scores can range from 0 to 56 with higher scores indicating higher perceived stress
Sleep quality - subjective | Day 1 (At-Home Session)
  Subjectively assessed by the Pittsburgh Sleep Quality Index (PQSI), which measures components of sleep: sleep duration, disturbance, sleep latency, daytime dysfunction due to sleepiness, sleep efficiency, overall sleep quality, and sleep medication use, with higher scores reflecting poorer sleep quality. From these 7 questions, a global score of 0 to 21 is created with higher values indicative of poorer sleep quality.
Sleep quantity and quality - device measured | Day 1 (At-Home Session)
  Measured via Garmin smartwatch for the total sleep duration and efficiency.
Physical activity | Day 1 (At-Home Session)
  Measured via Garmin smartwatch for time in moderate-vigorous physical activity, and step counts.
Sedentary time | Day 1 (At-Home Session)
  Measured via Garmin smartwatch for time spent sitting.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No